CLINICAL TRIAL: NCT01831466
Title: A Phase 2b, Multi-site, Randomized, Double-blind, Vehicle-controlled, Parallel-group Study Of The Efficacy, Safety, Local Tolerability And Pharmacokinetics Of 2 Dose Strengths And 2 Regimens Of Tofacitinib Ointment In Subjects With Chronic Plaque Psoriasis.
Brief Title: Tofacitinib Ointment For Chronic Plaque Psoriasis
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: A3921082; 2012-005645-20 (EudraCT Number)
Record Dates: First submitted 2013-03-28; First posted 2013-04-15 (Estimated); Results first posted 2015-11-25 (Estimated); Last update posted 2015-11-25 (Estimated); Status verified 2015-10

CONDITIONS: Psoriasis Vulgaris; Psoriasis
Keywords: plaque psoriasis; vulgaris; topical treatment; skin diseases; papulosquamous; Tofacitinib; CP-690550; Xeljanz; psoriasis; moderate; severe; itch; nail psoriasis
MeSH Terms: conditions — Psoriasis; Skin Diseases; Lymphoma, Follicular; Pruritus

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (6):
- Treatment Group A (Experimental)
  Interventions: Drug: tofacitinib ointment 20 mg/g
- Treatment Group B (Experimental)
  Interventions: Drug: tofacitinib ointment 10 mg/g
- Treatment Group C (Placebo Comparator)
  Interventions: Drug: placebo ointment (vehicle)
- Treatment Group D (Experimental)
  Interventions: Drug: tofacitinib ointment 20 mg/g
- Treatment Group E (Experimental)
  Interventions: Drug: tofacitinib ointment 10 mg/g
- Treatment Group F (Placebo Comparator)
  Interventions: Drug: placebo ointment (vehicle)

INTERVENTIONS:
Drug: tofacitinib ointment 20 mg/g — tofacitinib ointment 20 mg/g BID (twice daily) for 12 weeks
  Arms: Treatment Group A
Drug: tofacitinib ointment 10 mg/g — tofacitinib ointment 10 mg/g BID (twice daily) for 12 weeks
  Arms: Treatment Group B
Drug: placebo ointment (vehicle) — placebo ointment (vehicle) BID (twice daily) for 12 weeks
  Arms: Treatment Group C
Drug: tofacitinib ointment 20 mg/g — tofacitinib ointment 20 mg/g QD (once daily) for 12 weeks
  Arms: Treatment Group D
Drug: tofacitinib ointment 10 mg/g — tofacitinib ointment 10 mg/g QD (once daily) for 12 weeks
  Arms: Treatment Group E
Drug: placebo ointment (vehicle) — placebo ointment (vehicle) QD (once daily) for 12 weeks
  Arms: Treatment Group F

SUMMARY:
The study is beng done to test if tofacitinib ointment is safe and effective for people with plaque psoriasis. Two dose strengths of tofacitinib ointment (20 mg/g and 10 mg/g) applied once or twice daily are being tested. The safety and effectiveness of tofacitinib ointment used for 12 weeks will be compared to the safety and effectiveness of placebo ointment (vehicle) used for 12 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Have mild, moderate or severe plaque psoriasis (psoriasis vulgaris) for at least 6 months prior to Baseline
* At Baseline, have plaque psoriasis covering 2% to 20% of total body surface area (BSA) on the trunk and limbs (excluding palms, soles, and nails)
* If received certain treatments, should be off treatment for a minimum period of time (washout)

Exclusion Criteria:

* Currently have non-plaque forms of psoriasis or drug-induced psoriasis
* Require treatment with or cannot stop medication(s) prohibited during the study
* Have certain laboratory abnormalities at Baseline
* Current or history of certain infections
* Females who are pregnant, breastfeeding, or are of childbearing potential not using highly effective contraception

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 476 (Actual)
Dates: Start 2013-05; Primary Completion 2014-09 (Actual); Study Completion 2014-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (54):
- United States (29):
  - Burke Pharmaceutical Research, Hot Springs, Arkansas
  - Bakersfield Dermatology and Skin Cancer Medical Center, Bakersfield, California
  - UC Irvine Dermatology Research, Irvine, California
  - Dermatology Research Associates, Los Angeles, California
  - Park Avenue Dermatology, PA, Orange Park, Florida
  - Olympian Clinical Research, Tampa, Florida
  - Atlanta Dermatology, Vein & Research Center, Alpharetta, Georgia
  - Advanced Medical Research, Inc, Atlanta, Georgia
  - MedaPhase Inc., Newnan, Georgia
  - Dundee Dermatology, West Dundee, Illinois
  - Tufts Medical Center, Boston, Massachusetts
  - Massachusetts General Hospital - Clinical Unit for Research Trials in Skin (CURTIS), Boston, Massachusetts
  - Michigan Center for Skin Care Research, Clinton Township, Michigan
  - Dermatology Consulting Services, High Point, North Carolina
  - Wake Forest University Health Sciences, Winston-Salem, North Carolina
  - Radiant Research, Inc., Cincinnati, Ohio
  - Oregon Dermatology and Research Center, Portland, Oregon
  - Oregon Medical Research Center, PC, Portland, Oregon
  - Clinical Partners, LLC, Johnston, Rhode Island
  - Rhode Island Hospital, Providence, Rhode Island
  - Radiant Research, Inc., Greer, South Carolina
  - Health Concepts, Rapid City, South Dakota
  - Dermatology Research Associates, Nashville, Tennessee
  - Arlington Research Center Inc., Arlington, Texas
  - Dermatology Treatment and Research Center, Dallas, Texas
  - Menter Dermatology Research Institute, Dallas, Texas
  - Suzanne Bruce and Associates, PA, Houston, Texas
  - Lee Medical Associates, San Antonio, Texas
  - Progressive Clinical Research, San Antonio, Texas
- Canada (12):
  - Stratica Medical, Edmonton, Alberta
  - Dermadvances Research, Winnipeg, Manitoba
  - CCA Medical Research Corporation, Ajax, Ontario
  - Ultranova Skincare, Barrie, Ontario
  - Dermatrials Research, Hamilton, Ontario
  - The Guenther Dermatology Research Centre, London, Ontario
  - Lynderm Research Inc, Markham, Ontario
  - SKiN Centre for Dermatology, Peterborough, Ontario
  - K. Papp Clinical Research Inc., Waterloo, Ontario
  - XLR8 Medical Research, Windsor, Ontario
  - Innovaderm Research Inc, Montreal, Quebec
  - Siena Medical Research, Montreal, Quebec
- Denmark (2):
  - Dermatologisk Afdeling S, Aarhus C
  - Hudklinikken Herning, Herning
- Poland (11):
  - NZOZ Solumed, Poznan, Greater Poland Voivodeship
  - Klinika Ambroziak ESTEDERM Sp. z o.o.SKA, Warsaw, Masovian Voivodeship
  - Zdrowie Osteo-Medic s.c. Lidia i Artur Racewicz, Agnieszka i Jerzy Supronik, Bialystok
  - NZOZ Centrum Osteoporozy i Chorob Kostno-Stawowych J. Badurski Spolka Jawna, Bialystok
  - Pomorskie Centrum Traumatologii im.Mikolaja Kopernika w Gdansku Oddzial Dermatologii, Gdansk
  - Krakowskie Centrum Medyczne Sp. z o.o., Krakow
  - Maxxmed Centrum Zdrowia i Urody, Lublin
  - Gabinet Lekarski RTG USG Dr n. med. Pawel Skrzywanek; Pracownia Radiologiczna, Poznan
  - High-Med. Przychodnia Specjalistyczna, Warsaw
  - Wojskowy Instytut Medyczny, Warsaw
  - NZOZ multiMedica, Wroclaw

REFERENCES:
- [Derived] Papp KA, Bissonnette R, Gooderham M, Feldman SR, Iversen L, Soung J, Draelos Z, Mamolo C, Purohit V, Wang C, Ports WC. Treatment of plaque psoriasis with an ointment formulation of the Janus kinase inhibitor, tofacitinib: a Phase 2b randomized clinical trial. BMC Dermatol. 2016 Oct 3;16(1):15. doi: 10.1186/s12895-016-0051-4. PMID 27716172
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=A3921082&StudyName=Tofacitinib%20Ointment%20For%20Chronic%20Plaque%20Psoriasis

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants with mild (PGA-C score of 2), moderate (PGA-C score of 3), or severe (PGA-C score of 4) chronic plaque psoriasis were recruited for this study. The primary analysis population for this study included only the participants with mild and moderate disease.
Groups:
- Mild/Moderate: Tofacitinib 20 mg/Gram (mg/g) Twice Daily (BID): Participants with a baseline Calculated Physician's Global Assessment (PGA-C) score of mild (2) or moderate (3) applied tofacitinib ointment, 20 mg/g, BID for 12 weeks.
- Mild/Moderate: Tofacitinib 10 mg/g BID: Participants with a baseline PGA-C score of mild (2) or moderate (3) applied tofacitinib ointment, 10 mg/g, BID for 12 weeks.
- Mild/Moderate: Placebo (Vehicle) BID: Participants with a baseline PGA-C score of mild (2) or moderate (3) applied placebo ointment (vehicle), BID for 12 weeks.
- Mild/Moderate: Tofacitinib 20 mg/g Once Daily (QD): Participants with a baseline PGA-C score of mild (2) or moderate (3) applied tofacitinib ointment, 20 mg/g, QD for 12 weeks.
- Mild/Moderate: Tofacitinib 10 mg/g QD: Participants with a baseline PGA-C score of mild (2) or moderate (3) applied tofacitinib ointment 10 mg/g, QD for 12 weeks.
- Mild/Moderate: Placebo (Vehicle) QD: Participants with a baseline PGA-C score of mild (2) or moderate (3) applied placebo ointment (vehicle), QD for 12 weeks.
- Severe: Tofacitinib 20 mg/g BID: Participants with a baseline PGA-C score of severe (4) applied tofacitinib ointment, 20 mg/g, BID for 12 weeks.
- Severe: Tofacitinib 10 mg/g BID: Participants with a baseline PGA-C score of severe (4) applied tofacitinib ointment, 10 mg/g, BID for 12 weeks.
- Severe: Placebo (Vehicle) BID: Participants with a baseline PGA-C score of severe (4) applied placebo ointment (vehicle), BID for 12 weeks.
- Severe: Tofacitinib 20 mg/g QD: Participants with a baseline PGA-C score of severe (4) applied tofacitinib ointment, 20 mg/g, QD for 12 weeks.
- Severe: Tofacitinib 10 mg/g QD: Participants with a baseline PGA-C score of severe (4) applied tofacitinib ointment 10 mg/g, QD for 12 weeks.
- Severe: Placebo (Vehicle) QD: Participants with a baseline PGA-C score of severe (4) applied placebo ointment (vehicle), QD for 12 weeks.
Period: Overall Study
Arm/Group | Mild/Moderate: Tofacitinib 20 mg/Gram (mg/g) Twice Daily (BID) | Mild/Moderate: Tofacitinib 10 mg/g BID | Mild/Moderate: Placebo (Vehicle) BID | Mild/Moderate: Tofacitinib 20 mg/g Once Daily (QD) | Mild/Moderate: Tofacitinib 10 mg/g QD | Mild/Moderate: Placebo (Vehicle) QD | Severe: Tofacitinib 20 mg/g BID | Severe: Tofacitinib 10 mg/g BID | Severe: Placebo (Vehicle) BID | Severe: Tofacitinib 20 mg/g QD | Severe: Tofacitinib 10 mg/g QD | Severe: Placebo (Vehicle) QD
Started | 71 (Treated) | 70 (Treated) | 71 (Treated) | 70 (Treated) | 74 (Treated) | 74 (Treated) | 7 (Treated) | 7 (Treated) | 7 (Treated) | 7 (Treated) | 6 (Treated) | 7 (Treated)
Completed | 55 | 52 | 48 | 51 | 57 | 48 | 6 | 5 | 4 | 2 | 4 | 3
Not Completed | 16 | 18 | 23 | 19 | 17 | 26 | 1 | 2 | 3 | 5 | 2 | 4
Not completed — Protocol Violation | 1 | 1 | 2 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Other | 2 | 3 | 2 | 2 | 2 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Non-compliance with study treatment | 2 | 1 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Death | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Withdrawal by Subject | 6 | 3 | 3 | 3 | 3 | 5 | 0 | 0 | 0 | 1 | 0 | 1
Not completed — Lost to Follow-up | 0 | 1 | 4 | 2 | 0 | 3 | 0 | 0 | 0 | 1 | 0 | 1
Not completed — Lack of Efficacy | 5 | 8 | 7 | 6 | 9 | 8 | 1 | 1 | 2 | 2 | 2 | 0
Not completed — Adverse Event | 0 | 0 | 4 | 6 | 3 | 7 | 0 | 1 | 1 | 1 | 0 | 2

BASELINE CHARACTERISTICS:
Population: Full Analysis Set (FAS) - included all participants who were randomized to the study, received at least one dose of the randomized investigational drug (tofacitinib or vehicle), and were in a baseline PGA-C category of mild (2), moderate (3) or severe (4).
Groups:
- Mild/Moderate: Tofacitinib 20 mg/g BID: Participants with a baseline PGA-C score of mild (2) or moderate (3) applied tofacitinib ointment, 20 mg/g, BID for 12 weeks.
- Mild/Moderate: Tofacitinib 20 mg/g QD: Participants with a baseline PGA-C score of mild (2) or moderate (3) applied tofacitinib ointment, 20 mg/g, QD for 12 weeks.
- Total: Total of all reporting groups
Arm/Group | Mild/Moderate: Tofacitinib 20 mg/g BID | Mild/Moderate: Tofacitinib 10 mg/g BID | Mild/Moderate: Placebo (Vehicle) BID | Mild/Moderate: Tofacitinib 20 mg/g QD | Mild/Moderate: Tofacitinib 10 mg/g QD | Mild/Moderate: Placebo (Vehicle) QD | Severe: Tofacitinib 20 mg/g BID | Severe: Tofacitinib 10 mg/g BID | Severe: Placebo (Vehicle) BID | Severe: Tofacitinib 20 mg/g QD | Severe: Tofacitinib 10 mg/g QD | Severe: Placebo (Vehicle) QD | Total
Number analyzed (Participants) | 71 | 70 | 71 | 70 | 74 | 74 | 7 | 7 | 7 | 7 | 6 | 7 | 471
Age, Customized [Number; unit: Participants]
  < 18 years | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  18-44 years | 30 | 23 | 25 | 21 | 30 | 25 | 2 | 0 | 1 | 3 | 3 | 2 | 165
  45-64 years | 28 | 34 | 34 | 38 | 35 | 39 | 4 | 6 | 4 | 2 | 2 | 2 | 228
  >= 65 years | 13 | 13 | 12 | 11 | 9 | 10 | 1 | 1 | 2 | 2 | 1 | 3 | 78
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 28 | 23 | 30 | 33 | 24 | 32 | 1 | 3 | 1 | 1 | 0 | 0 | 176
  Male | 43 | 47 | 41 | 37 | 50 | 42 | 6 | 4 | 6 | 6 | 6 | 7 | 295

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants Achieving a PGA-C Response of Clear (0) or Almost Clear (1) and Greater Than or Equal to (≥) 2 Grade/Point Improvement From Baseline at Week 12
Description: Clinical signs of plaque psoriasis (erythema [E], induration [I], and scaling [S]) were scored separately according to a 5-point severity scale (0 to 4) to provide PGA subscores, which described the overall severity of each clinical sign. The PGA-C was a static assessment; i.e., without regard to a previous assessment. The PGA subscores are then summed and averaged after which the total average was rounded to the nearest whole number to determine the PGA-C score and category. A higher score indicated a higher level of severity. 0 is equal to (=) cleared except for any residual discoloration and 1=almost clear, majority of lesions had individual scores for E+I+S that when summed, averaged, and rounded equaled 1.
Time Frame: Baseline, Week 12
Population: The mild/moderate full analysis set (FASm) included all participants in the FAS with a baseline PGA-C disease severity of mild (2) or moderate (3). A participant with a missing value was considered a non-responder.
Measure: Number; unit: Percentage of Participants
Arm/Group | Mild/Moderate: Tofacitinib 20 mg/g BID | Mild/Moderate: Tofacitinib 10 mg/g BID | Mild/Moderate: Placebo (Vehicle) BID | Mild/Moderate: Tofacitinib 20 mg/g QD | Mild/Moderate: Tofacitinib 10 mg/g QD | Mild/Moderate: Placebo (Vehicle) QD
Number analyzed (Participants) | 71 | 70 | 71 | 70 | 74 | 74
Percentage of Participants | 21.1 | 12.9 | 16.9 | 20.0 | 21.6 | 17.6
Statistical Analysis 1: Comparison: Mild/Moderate: Tofacitinib 20 mg/g BID vs Mild/Moderate: Placebo (Vehicle) BID; Test type: Superiority or Other; p = 0.5425, Cochran-Mantel-Haenszel; Difference in response rates = 3.9, 80% CI 2-sided [-4.3 to 12.0], Standard Error of Mean 6.36
Statistical Analysis 2: Comparison: Mild/Moderate: Tofacitinib 10 mg/g BID vs Mild/Moderate: Placebo (Vehicle) BID; Test type: Superiority or Other; p = 0.4976, Cochran-Mantel-Haenszel; Difference in response rates = -4.0, 80% CI 2-sided [-11.5 to 3.5], Standard Error of Mean 5.87
Statistical Analysis 3: Comparison: Mild/Moderate: Tofacitinib 20 mg/g QD vs Mild/Moderate: Placebo (Vehicle) QD; Test type: Superiority or Other; p = 0.6039, Cochran-Mantel-Haenszel; Difference in response rates = 3.3, 80% CI 2-sided [-4.9 to 11.5], Standard Error of Mean 6.36
Statistical Analysis 4: Comparison: Mild/Moderate: Tofacitinib 10 mg/g QD vs Mild/Moderate: Placebo (Vehicle) QD; Test type: Superiority or Other; p = 0.5279, Cochran-Mantel-Haenszel; Difference in response rate = 4.0, 80% CI 2-sided [-4.1 to 12.1], Standard Error of Mean 6.34

2. Primary Outcome: Percentage of Participants Achieving a PGA-C Response of Clear (0) or Almost Clear (1) and ≥2 Grade/Point Improvement From Baseline at Week 8
Description: Clinical signs of plaque psoriasis (E, I, and S) were scored separately according to a 5-point severity scale (0 to 4) to provide PGA subscores, which described the overall severity of each clinical sign. The PGA-C was a static assessment; i.e., without regard to a previous assessment. The PGA subscores are then summed and averaged after which the total average was rounded to the nearest whole number to determine the PGA-C score and category. A higher score indicated a higher level of severity. 0 is equal to (=) cleared except for any residual discoloration and 1=almost clear, majority of lesions had individual scores for E+I+S that when summed, averaged, and rounded equaled 1.
Time Frame: Baseline, Week 8
Population: FASm. A participant with a missing value was considered a non-responder.
Measure: Number; unit: Percentage of Participants
Arm/Group | Mild/Moderate: Tofacitinib 20 mg/g BID | Mild/Moderate: Tofacitinib 10 mg/g BID | Mild/Moderate: Placebo (Vehicle) BID | Mild/Moderate: Tofacitinib 20 mg/g QD | Mild/Moderate: Tofacitinib 10 mg/g QD | Mild/Moderate: Placebo (Vehicle) QD
Number analyzed (Participants) | 71 | 70 | 71 | 70 | 74 | 74
Percentage of Participants | 22.5 | 10.0 | 11.3 | 18.6 | 14.9 | 8.1
Statistical Analysis 1: Comparison: Mild/Moderate: Tofacitinib 20 mg/g BID vs Mild/Moderate: Placebo (Vehicle) BID; Test type: Superiority or Other; p = 0.0710, Cochran-Mantel-Haenszel; Difference in response rates = 10.8, 80% CI 2-sided [3.1 to 18.5], Standard Error of Mean 5.99
Statistical Analysis 2: Comparison: Mild/Moderate: Tofacitinib 10 mg/g BID vs Mild/Moderate: Placebo (Vehicle) BID; Test type: Superiority or Other; p = 0.8175, Cochran-Mantel-Haenszel; Difference in response rates = -1.2, 80% CI 2-sided [-7.9 to 5.5], Standard Error of Mean 5.20
Statistical Analysis 3: Comparison: Mild/Moderate: Tofacitinib 20 mg/g QD vs Mild/Moderate: Placebo (Vehicle) QD; Test type: Superiority or Other; p = 0.0513, Cochran-Mantel-Haenszel; Difference in response rates = 11.0, 80% CI 2-sided [3.8 to 18.2], Standard Error of Mean 5.63
Statistical Analysis 4: Comparison: Mild/Moderate: Tofacitinib 10 mg/g QD vs Mild/Moderate: Placebo (Vehicle) QD; Test type: Superiority or Other; p = 0.2021, Cochran-Mantel-Haenszel; Difference in response rates = 6.7, 80% CI 2-sided [-0.0 to 13.4], Standard Error of Mean 5.23

3. Secondary Outcome: Percentage of Participants Achieving a PGA-C Response of Clear (0) or Almost Clear (1) at Week 12
Description: as for outcome 2
Time Frame: Week 12
Population: FASm. A participant with a missing value was considered a non-responder.
Measure: Number; unit: Percentage of Participants
Arm/Group | Mild/Moderate: Tofacitinib 20 mg/g BID | Mild/Moderate: Tofacitinib 10 mg/g BID | Mild/Moderate: Placebo (Vehicle) BID | Mild/Moderate: Tofacitinib 20 mg/g QD | Mild/Moderate: Tofacitinib 10 mg/g QD | Mild/Moderate: Placebo (Vehicle) QD
Number analyzed (Participants) | 71 | 70 | 71 | 70 | 74 | 74
Percentage of Participants | 33.8 | 25.7 | 23.9 | 27.1 | 29.7 | 23.0

4. Secondary Outcome: Percentage of Participants Achieving a PGA-C Response of Clear (0) or Almost Clear (1) at Week 8
Description: as for outcome 2
Time Frame: Week 8
Population: FASm. A participant with a missing value was considered a non-responder.
Measure: Number; unit: Percentage of Participants
Arm/Group | Mild/Moderate: Tofacitinib 20 mg/g BID | Mild/Moderate: Tofacitinib 10 mg/g BID | Mild/Moderate: Placebo (Vehicle) BID | Mild/Moderate: Tofacitinib 20 mg/g QD | Mild/Moderate: Tofacitinib 10 mg/g QD | Mild/Moderate: Placebo (Vehicle) QD
Number analyzed (Participants) | 71 | 70 | 71 | 70 | 74 | 74
Percentage of Participants | 36.6 | 20.0 | 22.5 | 32.9 | 21.6 | 12.2

5. Secondary Outcome: Percentage of Participants Achieving a Gestalt Physician's Global Assessment (PGA-G) Response of Clear (0) or Almost Clear (1) and ≥2 Grade/Point Improvement From Baseline at Week 12
Description: Clinical signs of plaque psoriasis (E, I and S) were scored separately according to a 5-point severity scale (0 to 4) to provide PGA subscores, which described the overall severity of each clinical sign. After scoring each of the PGA subscores, a clinical evaluator of psoriasis performed an assessment of the overall severity of psoriasis and assigned a PGA-G score and category. 0=Clear, except for any residual discoloration (post-inflammatory hyperpigmentation and/or hypopigmentation) and 1=almost clear, the psoriasis is not entirely cleared and remaining plaques are light pink (not including post inflammatory hyperpigmentation), and/or have barely palpable elevation and/or have occasional fine scale. The PGA-G was a static assessment; i.e., without regard to a previous assessment.
Time Frame: Baseline, Week 12
Population: FASm. A participant with a missing value was considered a non-responder.
Measure: Number; unit: Percentage of Participants
Arm/Group | Mild/Moderate: Tofacitinib 20 mg/g BID | Mild/Moderate: Tofacitinib 10 mg/g BID | Mild/Moderate: Placebo (Vehicle) BID | Mild/Moderate: Tofacitinib 20 mg/g QD | Mild/Moderate: Tofacitinib 10 mg/g QD | Mild/Moderate: Placebo (Vehicle) QD
Number analyzed (Participants) | 71 | 70 | 71 | 70 | 74 | 74
Percentage of Participants | 18.3 | 11.4 | 14.1 | 15.7 | 18.9 | 12.2

6. Secondary Outcome: Percentage of Participants Achieving a PGA-G Response of Clear (0) or Almost Clear (1) and ≥2 Grade/Point Improvement From Baseline at Week 8
Description: as for outcome 5
Time Frame: Baseline, Week 8
Population: FASm. A participant with a missing value was considered a non-responder.
Measure: Number; unit: Percentage of Participants
Arm/Group | Mild/Moderate: Tofacitinib 20 mg/g BID | Mild/Moderate: Tofacitinib 10 mg/g BID | Mild/Moderate: Placebo (Vehicle) BID | Mild/Moderate: Tofacitinib 20 mg/g QD | Mild/Moderate: Tofacitinib 10 mg/g QD | Mild/Moderate: Placebo (Vehicle) QD
Number analyzed (Participants) | 71 | 70 | 71 | 70 | 74 | 74
Percentage of Participants | 21.1 | 7.1 | 11.3 | 15.7 | 9.5 | 4.1

7. Secondary Outcome: Percent Change From Baseline to Week 12 in Psoriasis Area and Severity Index (PASI)
Description: Combined assessment of lesion severity and area affected into single score. Body was divided into 4 regions: head, arms, trunk, legs. For each region, percent (%) area of skin involved was estimated: 0=0% to 6=90-100%. Severity was estimated by clinical signs: erythema, induration, scaling; scale: 0=none to 4=maximum. Final PASI = sum of severity parameters for each region*area score*weight of region (head: 0.1, arms: 0.2, body: 0.3, legs: 0.4); total possible score range: 0=no disease to 72=maximal disease. The maximum PASI score was <72 since the PASI assessment excluded scalp, palms, finger nails, soles, and toe nails.
Time Frame: Baseline, Week 12
Population: FASm. Only observed data were analyzed.
Measure: Mean (Standard Deviation); unit: Percent Change from Baseline
Arm/Group | Mild/Moderate: Tofacitinib 20 mg/g BID | Mild/Moderate: Tofacitinib 10 mg/g BID | Mild/Moderate: Placebo (Vehicle) BID | Mild/Moderate: Tofacitinib 20 mg/g QD | Mild/Moderate: Tofacitinib 10 mg/g QD | Mild/Moderate: Placebo (Vehicle) QD
Number analyzed (Participants) | 58 | 57 | 55 | 53 | 62 | 52
Percent Change from Baseline | -36.6 (40.88) | -35.7 (43.78) | -32.0 (49.47) | -38.6 (36.37) | -31.4 (42.36) | -30.0 (38.68)

8. Secondary Outcome: Percent Change From Baseline to Week 8 in PASI
Description: Combined assessment of lesion severity and area affected into single score. Body was divided into 4 regions: head, arms, trunk, legs. For each region, percent area of skin involved was estimated: 0=0% to 6=90-100%. Severity was estimated by clinical signs: erythema, induration, scaling; scale: 0=none to 4=maximum. Final PASI = sum of severity parameters for each region*area score*weight of region (head: 0.1, arms: 0.2, body: 0.3, legs: 0.4); total possible score range: 0=no disease to 72=maximal disease. The maximum PASI score was <72 since the PASI assessment excluded scalp, palms, finger nails, soles, and toe nails.
Time Frame: Baseline, Week 8
Population: FASm. Only observed data were analyzed.
Measure: Mean (Standard Deviation); unit: Percent Change from Baseline
Arm/Group | Mild/Moderate: Tofacitinib 20 mg/g BID | Mild/Moderate: Tofacitinib 10 mg/g BID | Mild/Moderate: Placebo (Vehicle) BID | Mild/Moderate: Tofacitinib 20 mg/g QD | Mild/Moderate: Tofacitinib 10 mg/g QD | Mild/Moderate: Placebo (Vehicle) QD
Number analyzed (Participants) | 61 | 64 | 55 | 60 | 67 | 58
Percent Change from Baseline | -36.7 (36.01) | -29.1 (40.86) | -28.8 (37.06) | -36.5 (33.87) | -29.0 (29.47) | -27.1 (32.93)

9. Secondary Outcome: Percentage of Participants Achieving at Least a 75% Reduction in PASI Response (PASI75), Relative to Baseline at Week 12
Description: as for outcome 8
Time Frame: Baseline, Week 12
Population: FASm. A participant with a missing value was considered a non-responder.
Measure: Number; unit: Percentage of Participants
Arm/Group | Mild/Moderate: Tofacitinib 20 mg/g BID | Mild/Moderate: Tofacitinib 10 mg/g BID | Mild/Moderate: Placebo (Vehicle) BID | Mild/Moderate: Tofacitinib 20 mg/g QD | Mild/Moderate: Tofacitinib 10 mg/g QD | Mild/Moderate: Placebo (Vehicle) QD
Number analyzed (Participants) | 71 | 70 | 71 | 70 | 74 | 74
Percentage of Participants | 16.9 | 12.9 | 12.7 | 15.7 | 10.8 | 6.8

10. Secondary Outcome: Percentage of Participants Achieving PASI75, Relative to Baseline at Week 8
Description: as for outcome 8
Time Frame: Baseline, Week 8
Population: FASm. A participant with a missing value was considered a non-responder.
Measure: Number; unit: Percentage of Participants
Arm/Group | Mild/Moderate: Tofacitinib 20 mg/g BID | Mild/Moderate: Tofacitinib 10 mg/g BID | Mild/Moderate: Placebo (Vehicle) BID | Mild/Moderate: Tofacitinib 20 mg/g QD | Mild/Moderate: Tofacitinib 10 mg/g QD | Mild/Moderate: Placebo (Vehicle) QD
Number analyzed (Participants) | 71 | 70 | 71 | 70 | 74 | 74
Percentage of Participants | 14.1 | 8.6 | 7.0 | 15.7 | 6.8 | 6.8

11. Secondary Outcome: Percent Change From Baseline to Week 12 in Body Surface Area (BSA) Affected With Psoriasis
Description: Assessment of BSA with psoriasis was performed separately for 4 body regions: head and neck, upper limbs, trunk (including axillae and groin), and lower limbs (including buttocks). The percent surface area with psoriasis was estimated by means of the handprint method, where the full palmar hand of the participant represents approximately 1% of the total BSA. The number of handprints of psoriatic skin in a body region can be used to determine the extent (%) to which a body regions is involved with psoriasis. BSA (%)=the sum of the BSAs of the 4 body regions. BSA assessment excluded head and neck, palms, finger nails, soles and toe nails.
Time Frame: Baseline, Week 12
Population: FASm. Only observed data were analyzed.
Measure: Mean (Standard Deviation); unit: Percent Change from Baseline
Arm/Group | Mild/Moderate: Tofacitinib 20 mg/g BID | Mild/Moderate: Tofacitinib 10 mg/g BID | Mild/Moderate: Placebo (Vehicle) BID | Mild/Moderate: Tofacitinib 20 mg/g QD | Mild/Moderate: Tofacitinib 10 mg/g QD | Mild/Moderate: Placebo (Vehicle) QD
Number analyzed (Participants) | 58 | 57 | 55 | 53 | 62 | 52
Percent Change from Baseline | -32.8 (40.92) | -27.5 (36.40) | -27.7 (43.43) | -24.6 (36.29) | -15.6 (36.63) | -11.2 (56.38)

12. Secondary Outcome: Percent Change From Baseline to Week 8 in BSA Affected With Psoriasis
Description: as for outcome 11
Time Frame: Baseline, Week 8
Population: FASm. Only observed data were analyzed.
Measure: Mean (Standard Deviation); unit: Percent Change from Baseline
Arm/Group | Mild/Moderate: Tofacitinib 20 mg/g BID | Mild/Moderate: Tofacitinib 10 mg/g BID | Mild/Moderate: Placebo (Vehicle) BID | Mild/Moderate: Tofacitinib 20 mg/g QD | Mild/Moderate: Tofacitinib 10 mg/g QD | Mild/Moderate: Placebo (Vehicle) QD
Number analyzed (Participants) | 61 | 64 | 55 | 60 | 67 | 58
Percent Change from Baseline | -25.4 (44.75) | -22.5 (35.87) | -20.5 (34.90) | -17.8 (28.59) | -9.0 (30.08) | -11.7 (38.29)

13. Secondary Outcome: Change From Baseline to Week 12 in Clinic-Based Itch Severity Item (ISI) Scores
Description: The severity of itch (pruritus) due to psoriasis was assessed using the ISI. Participants were asked to assess their "worst itching due to psoriasis over the past 24 hours" on a numeric rating scale anchored by the terms "no itching" (0) and "worst possible itching" (10) at the ends. Participants completed the ISI assessments at the clinic (i.e., clinic-based).
Time Frame: Baseline, Week 12
Population: FASm. Only observed data were analyzed.
Measure: Mean (Standard Deviation); unit: Score on a Scale
Arm/Group | Mild/Moderate: Tofacitinib 20 mg/g BID | Mild/Moderate: Tofacitinib 10 mg/g BID | Mild/Moderate: Placebo (Vehicle) BID | Mild/Moderate: Tofacitinib 20 mg/g QD | Mild/Moderate: Tofacitinib 10 mg/g QD | Mild/Moderate: Placebo (Vehicle) QD
Number analyzed (Participants) | 57 | 57 | 55 | 52 | 62 | 52
Score on a Scale | -2.88 (3.140) | -2.89 (3.320) | -1.73 (2.460) | -2.38 (3.182) | -1.94 (3.151) | -1.50 (2.961)

14. Secondary Outcome: Change From Baseline to Week 8 in Clinic-Based ISI Scores
Description: as for outcome 13
Time Frame: Baseline, Week 8
Population: FASm. Only observed data were analyzed.
Measure: Mean (Standard Deviation); unit: Score on a Scale
Arm/Group | Mild/Moderate: Tofacitinib 20 mg/g BID | Mild/Moderate: Tofacitinib 10 mg/g BID | Mild/Moderate: Placebo (Vehicle) BID | Mild/Moderate: Tofacitinib 20 mg/g QD | Mild/Moderate: Tofacitinib 10 mg/g QD | Mild/Moderate: Placebo (Vehicle) QD
Number analyzed (Participants) | 61 | 64 | 55 | 59 | 66 | 58
Score on a Scale | -3.07 (2.971) | -2.38 (2.984) | -1.45 (2.847) | -2.49 (2.769) | -1.91 (3.166) | -1.34 (3.285)

15. Secondary Outcome: Change From Baseline to Week 12 in the Dermatology Life Quality Index (DLQI) Total Score
Description: DLQI is the dermatology-specific quality of life measure used for psoriatic population. The 10-item questionnaire assesses participant health-related quality of life (daily activities, personal relationships, symptoms and feelings, leisure, work and school, and treatment). The DLQI questions are rated by the participant as 0 (not at all/not relevant) to 3 (very much) with a total score range of 0 (best) to 30 (worst); higher scores indicate poor quality of life.
Time Frame: Baseline, Week 12
Population: FASm. Only observed data were analyzed.
Measure: Mean (Standard Deviation); unit: Score on a Scale
Arm/Group | Mild/Moderate: Tofacitinib 20 mg/g BID | Mild/Moderate: Tofacitinib 10 mg/g BID | Mild/Moderate: Placebo (Vehicle) BID | Mild/Moderate: Tofacitinib 20 mg/g QD | Mild/Moderate: Tofacitinib 10 mg/g QD | Mild/Moderate: Placebo (Vehicle) QD
Number analyzed (Participants) | 58 | 57 | 55 | 53 | 62 | 52
Score on a Scale | -4.6 (5.55) | -3.2 (5.32) | -2.6 (5.45) | -5.6 (7.04) | -3.3 (5.97) | -2.3 (6.34)

16. Secondary Outcome: Change From Baseline to Week 8 in the DLQI Total Score
Description: as for outcome 15
Time Frame: Baseline, Week 8
Population: FASm. Only observed data were analyzed.
Measure: Mean (Standard Deviation); unit: Score on a Scale
Arm/Group | Mild/Moderate: Tofacitinib 20 mg/g BID | Mild/Moderate: Tofacitinib 10 mg/g BID | Mild/Moderate: Placebo (Vehicle) BID | Mild/Moderate: Tofacitinib 20 mg/g QD | Mild/Moderate: Tofacitinib 10 mg/g QD | Mild/Moderate: Placebo (Vehicle) QD
Number analyzed (Participants) | 61 | 64 | 55 | 60 | 67 | 58
Score on a Scale | -4.6 (5.16) | -2.6 (4.98) | -2.8 (4.01) | -5.0 (5.85) | -2.7 (4.79) | -2.2 (5.63)

17. Secondary Outcome: Percentage of Participants Achieving a Patient's Global Assessment (PtGA) Response of Clear (0) or Almost Clear (1) and ≥2 Grade/Point Improvement From Baseline at Week 12 for Participants With a PtGA Score ≥2 at Baseline
Description: The PtGA asks the participant to evaluate the overall cutaneous disease at that point in time on a single item, 5-point scale (0=clear; 1=almost clear; 2=mild; 3=moderate; 4=severe).
Time Frame: Baseline, Week 12
Population: FASm. Only observed data were analyzed.
Measure: Number; unit: Percentage of Participants
Arm/Group | Mild/Moderate: Tofacitinib 20 mg/g BID | Mild/Moderate: Tofacitinib 10 mg/g BID | Mild/Moderate: Placebo (Vehicle) BID | Mild/Moderate: Tofacitinib 20 mg/g QD | Mild/Moderate: Tofacitinib 10 mg/g QD | Mild/Moderate: Placebo (Vehicle) QD
Number analyzed (Participants) | 57 | 57 | 55 | 53 | 62 | 52
Percentage of Participants | 8.8 | 17.5 | 7.3 | 13.2 | 14.5 | 7.7

18. Secondary Outcome: Percentage of Participants Achieving a PtGA Response of Clear (0) or Almost Clear (1) and ≥2 Grade/Point Improvement From Baseline at Week 8 for Participants With a PtGA Score ≥2 at Baseline
Description: as for outcome 17
Time Frame: Baseline, Week 8
Population: FASm. Only observed data were analyzed.
Measure: Number; unit: Percentage of Participants
Arm/Group | Mild/Moderate: Tofacitinib 20 mg/g BID | Mild/Moderate: Tofacitinib 10 mg/g BID | Mild/Moderate: Placebo (Vehicle) BID | Mild/Moderate: Tofacitinib 20 mg/g QD | Mild/Moderate: Tofacitinib 10 mg/g QD | Mild/Moderate: Placebo (Vehicle) QD
Number analyzed (Participants) | 60 | 64 | 55 | 60 | 67 | 58
Percentage of Participants | 5.0 | 6.3 | 10.9 | 10.0 | 6.0 | 1.7

ADVERSE EVENTS:
Time Frame: SAEs were assessed from informed consent through and including 28 calendar days after last administration of study treatment. Non-SAEs were recorded from time of first dose of study treatment through last participant visit.
Description: The same event may appear as both an AE and an SAE. However, what is presented are distinct events. An event may be categorized as serious in 1 participant and as nonserious in another participant, or 1 participant may have experienced both a serious and nonserious event during the study. All AEs (including treatment area AEs) are presented.
Arm/Group | Mild/Moderate: Tofacitinib 20 mg/g BID | Mild/Moderate: Tofacitinib 10 mg/g BID | Mild/Moderate: Placebo (Vehicle) BID | Mild/Moderate: Tofacitinib 20 mg/g QD | Mild/Moderate: Tofacitinib 10 mg/g QD | Mild/Moderate: Placebo (Vehicle) QD | Severe: Tofacitinib 20 mg/g BID | Severe: Tofacitinib 10 mg/g BID | Severe: Placebo (Vehicle) BID | Severe: Tofacitinib 20 mg/g QD | Severe: Tofacitinib 10 mg/g QD | Severe: Placebo (Vehicle) QD
Serious Adverse Events (participants affected / at risk) | 0/71 | 5/70 | 2/71 | 0/70 | 2/74 | 1/74 | 0/7 | 0/7 | 0/7 | 0/7 | 0/6 | 1/7
Other Adverse Events (participants affected / at risk) | 30/71 | 29/70 | 27/71 | 34/70 | 28/74 | 40/74 | 2/7 | 4/7 | 4/7 | 3/7 | 2/6 | 2/7
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Mild/Moderate: Tofacitinib 20 mg/g BID (N=71) | Mild/Moderate: Tofacitinib 10 mg/g BID (N=70) | Mild/Moderate: Placebo (Vehicle) BID (N=71) | Mild/Moderate: Tofacitinib 20 mg/g QD (N=70) | Mild/Moderate: Tofacitinib 10 mg/g QD (N=74) | Mild/Moderate: Placebo (Vehicle) QD (N=74) | Severe: Tofacitinib 20 mg/g BID (N=7) | Severe: Tofacitinib 10 mg/g BID (N=7) | Severe: Placebo (Vehicle) BID (N=7) | Severe: Tofacitinib 20 mg/g QD (N=7) | Severe: Tofacitinib 10 mg/g QD (N=6) | Severe: Placebo (Vehicle) QD (N=7)
Arrhythmia (Cardiac disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Atrial fibrillation (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Cardiac failure congestive (Cardiac disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Myocardial infarction (Cardiac disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Non-cardiac chest pain (General disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Systemic inflammatory response syndrome (General disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Urinary tract infection (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Abdominal wound dehiscence (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Diabetes mellitus (Metabolism and nutrition disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Psoriatic arthropathy (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Transient ischaemic attack (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Mild/Moderate: Tofacitinib 20 mg/g BID (N=71) | Mild/Moderate: Tofacitinib 10 mg/g BID (N=70) | Mild/Moderate: Placebo (Vehicle) BID (N=71) | Mild/Moderate: Tofacitinib 20 mg/g QD (N=70) | Mild/Moderate: Tofacitinib 10 mg/g QD (N=74) | Mild/Moderate: Placebo (Vehicle) QD (N=74) | Severe: Tofacitinib 20 mg/g BID (N=7) | Severe: Tofacitinib 10 mg/g BID (N=7) | Severe: Placebo (Vehicle) BID (N=7) | Severe: Tofacitinib 20 mg/g QD (N=7) | Severe: Tofacitinib 10 mg/g QD (N=6) | Severe: Placebo (Vehicle) QD (N=7)
Anaemia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Leukocytosis (Blood and lymphatic system disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Leukopenia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Pancytopenia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Cerumen impaction (Ear and labyrinth disorders) | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Ear discomfort (Ear and labyrinth disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Vertigo (Ear and labyrinth disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Erythema of eyelid (Eye disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Eyelid oedema (Eye disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Lacrimation increased (Eye disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Abdominal pain upper (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Chronic gastritis (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Dental caries (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Diarrhoea (Gastrointestinal disorders) | 2 | 0 | 1 | 3 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Dyspepsia (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Food poisoning (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Gastritis (Gastrointestinal disorders) | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Hiatus hernia (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Inguinal hernia (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Nausea (Gastrointestinal disorders) | 2 | 1 | 1 | 1 | 3 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Tongue ulceration (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Vomiting (Gastrointestinal disorders) | 0 | 0 | 1 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Application site pain (General disorders) | 0 | 0 | 1 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0
Application site papules (General disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Asthenia (General disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Chest pain (General disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Fatigue (General disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Influenza like illness (General disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Oedema peripheral (General disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Pyrexia (General disorders) | 0 | 0 | 1 | 1 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Seasonal allergy (Immune system disorders) | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Bacteriuria (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Bronchitis (Infections and infestations) | 2 | 1 | 0 | 1 | 1 | 1 | 1 | 0 | 1 | 0 | 0 | 0
Chronic tonsillitis (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Conjunctivitis (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Ear infection (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Fungal infection (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Gastroenteritis viral (Infections and infestations) | 0 | 0 | 0 | 2 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Gastrointestinal viral infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Gingivitis (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Infected bites (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Influenza (Infections and infestations) | 0 | 0 | 1 | 2 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Nasopharyngitis (Infections and infestations) | 3 | 2 | 1 | 5 | 7 | 11 | 0 | 1 | 0 | 0 | 0 | 0
Oral candidiasis (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Oral herpes (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Otitis externa (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Paronychia (Infections and infestations) | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Pharyngitis (Infections and infestations) | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Pulpitis dental (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Pyelonephritis (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Rash pustular (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Rhinitis (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Sepsis (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Sinusitis (Infections and infestations) | 1 | 1 | 2 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Tooth abscess (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Tooth infection (Infections and infestations) | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Upper respiratory tract infection (Infections and infestations) | 2 | 10 | 6 | 2 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0
Urinary tract infection (Infections and infestations) | 0 | 2 | 6 | 1 | 2 | 1 | 0 | 0 | 0 | 1 | 0 | 0
Viral upper respiratory tract infection (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Accident at work (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Arthropod bite (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Burns first degree (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Drug dispensing error (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Fall (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Foot fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Laceration (Injury, poisoning and procedural complications) | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Muscle strain (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 1 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Post-traumatic neck syndrome (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Procedural pain (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Scar (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Skin abrasion (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Alanine aminotransferase increased (Investigations) | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Aspartate aminotransferase increased (Investigations) | 0 | 2 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Blood cholesterol increased (Investigations) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Blood creatinine increased (Investigations) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Blood triglycerides increased (Investigations) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Eosinophil percentage increased (Investigations) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Gamma-glutamyltransferase increased (Investigations) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Liver function test abnormal (Investigations) | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Low density lipoprotein increased (Investigations) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Vitamin B12 decreased (Investigations) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
White blood cell count decreased (Investigations) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Dehydration (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Hypercholesterolaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 1 | 2 | 0 | 0 | 0 | 0 | 0 | 0
Hyperglycaemia (Metabolism and nutrition disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1
Hyperlipidaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Hypertriglyceridaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Hypoglycaemia (Metabolism and nutrition disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Hypokalaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Hypomagnesaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Type 2 diabetes mellitus (Metabolism and nutrition disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Exostosis (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Joint range of motion decreased (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Joint stiffness (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Neck pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Psoriatic arthropathy (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 1 | 1 | 2 | 0 | 0 | 0 | 0 | 0 | 0
Spinal osteoarthritis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Squamous cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Dizziness (Nervous system disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0
Dysaesthesia (Nervous system disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Generalised tonic-clonic seizure (Nervous system disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Headache (Nervous system disorders) | 0 | 2 | 2 | 3 | 3 | 2 | 0 | 0 | 0 | 0 | 0 | 0
Migraine (Nervous system disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Tension headache (Nervous system disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Anxiety (Psychiatric disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Depression (Psychiatric disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Insomnia (Psychiatric disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Stress (Psychiatric disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Haematuria (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Nephrolithiasis (Renal and urinary disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Proteinuria (Renal and urinary disorders) | 0 | 0 | 0 | 1 | 1 | 2 | 0 | 0 | 0 | 0 | 0 | 0
Erectile dysfunction (Reproductive system and breast disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Asthma (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Catarrh (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Dry throat (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 2 | 0 | 3 | 0 | 0 | 0 | 0 | 0 | 0
Paranasal sinus discomfort (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Respiratory tract congestion (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Sinus congestion (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Sneezing (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Acne (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Dermal cyst (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Dermatitis contact (Skin and subcutaneous tissue disorders) | 1 | 1 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Dry skin (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0
Erythema (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Intertrigo (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Nail psoriasis (Skin and subcutaneous tissue disorders) | 2 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Onychoclasis (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Pruritus (Skin and subcutaneous tissue disorders) | 1 | 0 | 1 | 2 | 2 | 4 | 0 | 0 | 1 | 0 | 0 | 0
Psoriasis (Skin and subcutaneous tissue disorders) | 1 | 1 | 0 | 7 | 6 | 6 | 1 | 0 | 0 | 2 | 0 | 1
Rash macular (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Skin burning sensation (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Skin fissures (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Skin lesion (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Haematoma (Vascular disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Hypertension (Vascular disorders) | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Hypotension (Vascular disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Vasculitis (Vascular disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Hypothyroidism (Endocrine disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Abdominal tenderness (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Constipation (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Application site pruritus (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Cystitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Cystitis escherichia (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Erysipelas (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Impetigo (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Intervertebral disc degeneration (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Lipoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Glycosuria (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Vaginal haemorrhage (Reproductive system and breast disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

LIMITATIONS AND CAVEATS:
Efficacy results for participants in the severe population were not reported since this was considered an exploratory population.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The sponsor can review results communications prior to public release and can embargo communications regarding trial results for a period that is less than or equal to 60 days from the time submitted to the sponsor for review. The PI must remove any previously undisclosed Confidential Information (other than the Study results themselves) before public release.